CLINICAL TRIAL: NCT05921448
Title: In-depth Immunological Analysis of Airway Immunity Following Nasal Live Attenuated and Intramuscular Influenza Vaccine
Brief Title: Vaccine Pandemic Preparedness Through Airway Immunology Characterization
Acronym: VAXXAIR
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chronic Obstructive Pulmonary Disease Trial Network, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAXXAIR
Record Dates: First submitted 2023-06-18; First posted 2023-06-27 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Intervention Model Description: 2-arm randomized, placebo-controlled, multicenter, parallel group intervention study in patients aged between 18-49.
  Participants will be randomly allocated to one of four treatment groups.
  Conducted in adherence with Good Clinical Practice (GCP).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) . Encryption will be through a website (REDCap).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaxigripetra (Experimental): This arm will receive 1 dose of 0.5 mL Vaxigripetra (intra-muscular injection) and 1 dose of 0.2 mL placebo (nasal, 1 spray in each nostril).
  Interventions: Biological: Vaxigripetra
- Flumist (Experimental): 1 dose of 0.2 mL Flumist (nasal, 1 spray in each nostril) and 1 dose of 0.5 mL placebo (intra-muscular injection).
  Interventions: Biological: Flumist

INTERVENTIONS:
Biological: Vaxigripetra — Tetravalent intramuscular vaccine. Mechanism of action: The vaccine induces an immune reaction involving antibody production.
  Arms: Vaxigripetra
Biological: Flumist — Tetravalent live attenuated influenza vaccine administered as a nasal spray. Mechanism of action: Not fully understood according to the prescribing information, but may involve influenza-specific T-cells and antibodies (serum and mucosal).
  Arms: Flumist

SUMMARY:
The study aims to compare the effectiveness of live attenuated influenza vaccines (LAIV) and intramuscular-inactivated vaccines (IIV) in healthy individuals aged 18-49. It will investigate cellular and humoral responses, identify immunological markers for targeted vaccine improvement, and establish a collaborative platform for accelerated immunological and clinical vaccine research.

DETAILED DESCRIPTION:
There are several types of vaccines and the focus on the important role of vaccines in health has increased after the SARS-CoV-2 pandemic. Therefore, it is desired to investigate whether so-called 'live attenuated influenza vaccines' (LAIV) can prove more effective than the most frequently used 'intramuscular-inactivated vaccines' (IIV).

Several studies have previously compared the humoral and cellular response to LAIV and IIV and some of these have shown that LAIV elicits a more robust cellular response than intramuscularly administered vaccines.

In the study, the immunological differences in cellular and humoral response following vaccination either intramuscularly or nasally will be characterized. The patient group will consist of healthy individuals between 18-49 years of age. It is further desired to identify immunological markers that vaccines can be directed against in order to improve the immunological response. Finally, a platform for collaboration on accelerated immunological and clinical vaccine research will be established.

The study is a randomized, double-blind, placebo-controlled study. It is carried out in several locations and is Good Clinical Practice monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals (Charlson´s co-morbidity index :0, and investigator judged as healthy)
2. Age: 18-49 years
3. Total IgG levels in normal range (discretion of investigator according to local lab)
4. Total IgA levels (discretion of investigator according to local lab)
5. Undetectable HAI titres to the H3N2 component of the vaccines*
6. Normal CD4+ and CD8+ T-cell and normal B-cell counts
7. Reference levels from ISO-15189 accredited T-, B- and NK-cell count routine analyses will be applied.

   * If <20% of the first 100 screened persons apply to this criterion, this will be changed to a specific cut off based on the lowest quartile level of HAI titres to the H3N2 component of these 100 screened persons.

Exclusion Criteria:

1. Laboratory-confirmed influenza infection during the past year documented by a positive PCR test in the Danish Microbiological database or anamnestic reported influenza infection in the same period
2. Active smoker
3. BMI > 35 kg/m2
4. Women of childbearing potential not using safe contraception, or who are pregnant, or breast-feeding
5. Any allergies to components of or contraindication for Vaxigriptetra® or Flumist® incl. previous severe adverse reactions to influenza vaccinations or components of the vaccines
6. Use of immunosuppressive drugs* within the past 6 months or who are currently using them
7. HIV, HBV, HCV laboratory confirmed active infection at screening visit
8. Have an acute illness, including an oral temperature ≥ 38°C, within 3 days prior to vaccination
9. Have received any vaccines, including live-attenuated vaccines within 4 weeks before inclusion, or plan receipt of such vaccines within 30 days following the inclusion
10. Any known malignant neoplasm within 5 years (except basal carcinoma of the skin).
11. Severe mental illness or linguistic issues which significantly impedes cooperation
12. Inability to provide written informed consent

    * defined as: Azathioprin, methotrexate, cyclophosphamide, basiliximab, belimumab, anifrolumab, alemtuzumab, rituximab, mycophenolat, calcineurin inhibitors (ciclosporin, voclosporin and tacrolimus), mTOR inhibitors (everolimus and sirolimus), prednisolone (or any corticosteroid in doses above the equivalent of 5 mg prednisolone), TNF-α inhibitors (such as infliximab), anti-thymocyte globulin.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Day 28, mucosal immunity in nasopharynx (humoral) | Day -14 (baseline) [+/-5 days] vs. day +28 [+/-5 days]
  Time point: Comparison between day -14 (baseline) [+/-5 days] vs. day +28 [+/-5 days].
  Explanation: all individuals who have a ≥-4-fold rise in (A (H3N2) haemagglutinin vaccine-specific IgA in nasopharyngeal secretions will be characterized as outcome 1. All other individuals will be characterized as outcome 0.
  Material: Nasopharyngeal secretions Explanation: all individuals who have a ≥-4-fold rise in (A (H3N2) haemagglutinin vaccine-specific IgA in nasal secretions will be characterized as outcome 1. All other individuals will be characterized as outcome 0.
  Material: nasopharyngeal secretion.

SECONDARY OUTCOMES:
Day 7, mucosal immunity in nasopharynx (humoral) | Day -14 (baseline) [+/-5 days] vs. day +7 [+/-1 days]
  Time point: Comparison between day -14 (baseline) [+/-5 days] vs. day +7 [+/-1 days].
  Explanation: all individuals who have a ≥-4-fold rise in (A (H3N2) haemagglutinin vaccine-specific IgA in nasopharyngeal secretions will be characterized as outcome 1. All other individuals will be characterized as outcome 0.
  Material: Nasopharyngeal secretions Explanation: all individuals who have a ≥-4-fold rise in (A (H3N2) haemagglutinin vaccine-specific IgA in nasopharyngeal secretions will be characterized as outcome 1. All other individuals will be characterized as outcome 0.
  Material: Nasopharyngeal secretions Explanation: all individuals who have a ≥-4-fold rise in (A (H3N2)) haemagglutinin vaccine-specific IgA in nasal secretions will be characterized as outcome 1. All other individuals will be characterized as outcome 0.
  Material: nasopharyngeal secretion.
Day 28, mucosal immunity in Lower Airways (BALF) (humoral) | Day -14 (baseline) [+/-5 days] vs. day +28 [+/-5 days]
  Time point: Comparison between day -14 (baseline) [+/-5 days] vs. day +28 [+/-5 days].
  Explanation: all individuals who have a ≥-4-fold rise in (A (H3N2) haemagglutinin vaccine-specific IgA in nasopharyngeal secretions will be characterized as outcome 1. All other will be characterized as outcome 0.
Day 7, mucosal immunity in Lower Airways (BALF) (humoral) | Day -14 (baseline) [+/-5 days] vs. day +7 [+/-1 days]
  Time point: Comparison between day -14 (baseline) [+/-5 days] vs. day +7 [+/-1 days].
  Explanation: all individuals who have a ≥-4-fold rise in (A (H3N2) haemagglutinin vaccine-specific IgA in BALF will be characterized as outcome 1. All other individuals will be characterized as outcome 0.
Rise in mucosal antibody titre (humoral) | Day +28 [+/- 5 days]
  Hypothesis: Intranasally administered LAIV influenza vaccine will more often produce a ≥-4-fold rise in mucosal antibody titre against each of the remaining (non-H3N2) vaccine virus haemagglutinin antigens vaccine-specific antibody (IgG (when BALF) and IgA (when nasopharyngeal)) titres in respiratory secretions compared to intramuscular IIV tetravalent influenza vaccine.
  Time points: Day -14 (baseline), and i) day 28 [+/-5 days] ii) and day 7 [+/-1 day] after vaccination.
  Antigens: 1) A (H1N1) ; 2) B/Austria/1359417/2021 ; 3) B/Phuket/3073/2013 Material: BALF and nasopharyngeal secretion
Lower airways mucosal immunity, CD4+ (cellular) | Day -14 (baseline) vs. day +7
  Hypothesis: Intranasally administered LAIV influenza vaccine will lead to a higher number of Antigen activated* CD4+ T-lymphocytes in BALF measured at day -14 (baseline) vs. day +7 as compared to intramuscular IIV tetravalent influenza vaccine.
  Explanation: Fractions of CD4+ T-lymphocytes, that are antigen activated against an antigen pool composed of the antigens in the two utilized vaccines, will be measured at day -14 (baseline) and day +7.
  Fold changes will be compared between vaccine arms. Material: BALF.
  * A (H1N1) - A (H3N2) • B/Austria/1359417/2021 • B/Phuket/3073/2013
Systemic immunity (blood) (cellular) | Day -14 (baseline) vs. day +7
  Hypothesis: Intranasally administered LAIV influenza vaccine will lead to a higher number of Antigen activated* CD4+ T-lymphocytes in blood measured at day -14 (baseline) vs. day +7 as compared to intramuscular IIV tetravalent influenza vaccine.
  Explanation: Fractions of CD4+ T-lymphocytes, that are antigen activated against an antigen pool composed of the antigens in the two utilized vaccines, will be measured at day -14 (baseline) and day +7.
  Fold changes will be compared between vaccine arms. Material: Blood
  * A (H1N1) - A (H3N2) • B/Austria/1359417/2021 • B/Phuket/3073/2013

OTHER OUTCOMES:
Early changes in local immune profiles (cellular) | Day -14 (baseline) vs. day +7
  Hypothesis and explanation: Airway-delivered LAIV vaccine (Flumist) will induce early antigen specific T- lymphocytes as well as resident memory T- and B-cells locally in the respiratory tract that is characterized by activated TRM and TFH in BALF and mediastinal lymph nodes, and with higher levels of CXCR3pos-B-cells and BRM in BALF and respiratory mucosal tissue and mediatinal lymph nodes compared to that of intramuscular delivered trivalent flu vaccine.
  Material: BALF
Upper airways lymph node (Tonsil) immunity (cellular) | Day -14 (baseline) vs. day +7
  Hypothesis: Intranasally administered LAIV influenza vaccine will lead to a higher number of Antigen activated* CD4+ T-lymphocytes in lymphoid tissue from tonsils measured at day -14 (baseline) vs. day +7 as compared to intramuscular IIV tetravalent influenza vaccine.
  Explanation: Fractions of CD4+ and CD8+ T-lymphocytes, that are antigen activated against an antigen pool composed of the antigens in the two utilized vaccines, will be compared between day -14 (baseline) and day +7.
  Material: Lymphoid tissue from tonsils. Analysis of this hypothesis depends on feasibility (enough material)
  * A (H1N1) - A (H3N2) • B/Austria/1359417/2021 • B/Phuket/3073/2013
Lower airways mucosal immunity, CD8+ (cellular) | Day -14 (baseline) vs. day +7
  Hypothesis: Intranasally administered LAIV influenza vaccine will lead to a higher number of Antigen activated* CD8+ T-lymphocytes in BALF measured at day -14 (baseline) vs. day +7 as compared to intramuscular IIV tetravalent influenza vaccine.
  Explanation: Fractions of CD8+ T-lymphocytes, that are antigen activated against an antigen pool composed of the antigens in the two utilized vaccines, will be measured at day -14 (baseline) and day +7.
  Fold changes will be compared between vaccine arms. Material: BALF.
  * A (H1N1) - A (H3N2) • B/Austria/1359417/2021 • B/Phuket/3073/2013
Further exploratory humoral characterization | Day -14 (baseline), day +7 day +28 [+/-5 days], day +90 and day 180 [+/-5 days]
  Haemagglutinin antigens vaccine-specific antibody (IgG) titres in serum (HAI). This will be analysed in the following analyses:
  A. Number of participants with ≥-4-fold rise in serum antibody titres against each vaccine virus* B. Categorical and scalar associations between vaccine virus shedding (measured at days +1, +3, and +7 post-vaccination) and cellular and humoral immune responses.
  C. Proportion of study enrolled subjects achieving a HAI titre of ≥1:40 measured using antibody titre measured at -14 (baseline), day +7 day +28 [+/-5 days], day +90 and day 180 [+/-5 days] after vaccination.
  * A (H1N1) - A (H3N2) • B/Austria/1359417/2021 • B/Phuket/3073/2013

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Ulrik Stæhr Jensen, MD, PhD, Principal Investigator — Chronic Obstructive Pulmonary Disease Trial Network, Denmark
Locations (7):
- Denmark (6):
  - Copenhagen Hospital Biobank Unit, Department of Clinical Immunology, Rigshospitalet, Denmark, Copenhagen, Copenhagen
  - Diagnostic Immunology, Department of Clinical Immunology, Rigshospitalet, Denmark, Copenhagen, Copenhagen
  - Institute for Immunology and Microbiology (ISIM), Panum Institute, University of Copenhagen, Copenhagen, Copenhagen
  - Department of Medicine, Section of Respiratory Medicine, Herlev and Gentofte Hospital, Gentofte Municipality, Copenhagen
  - National Influenza Center for WHO at Statens Serum Institut (SSI), Copenhagen
  - Technical University of Denmark (DTU), Kongens Lyngby
- Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This has not yet been decided.